CLINICAL TRIAL: NCT06349200
Title: Comparing Binaural Beats and 432Hz Music for Reduction of Preoperative Anxiety in Root Canal Patients: an RCT Study
Brief Title: Comparing Binaural Beats and 432Hz Music for Reduction of Preoperative Anxiety in Root Canal Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Hafsa Zaki, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3197
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Dental Anxiety
Keywords: Preoperative Dental Anxiety; 432 Hz Music; Binaural Beats; White Noise; Audio Distraction; Root canal treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 432 Hz Music (Experimental): Group A will listen to music tuned to 432 Hz (Summer by Stefano Crespan Shantam on Spotify) using wireless headphones for 10 minutes.
  Interventions: Behavioral: 432 Hz music
- Binaural Beats (Experimental): Group B will listen to binaural beats (220 Hz for the right ear and 210 Hz for the left ear) using wireless headphones for 10 minutes. The frequencies will be generated by the mobile application BrainWaves Binaural Beats, MynioTech Apps, Chanpeco, Santa Catarina, Brazil.
  Interventions: Behavioral: Binaural beats
- Control (Active Comparator): Group C will be the active control group. The patients will listen to white noise for 10 minutes using wireless headphones.
  Interventions: Behavioral: White noise

INTERVENTIONS:
Behavioral: 432 Hz music — Music tuned to the 432 Hz frequency, as compared with other frequencies, has the advantage of providing utter calm, pleasure, and peace to its listeners. It has proven to be effective for reducing stress and improving sleep quality
  Other Names: Natural frequency music
  Arms: 432 Hz Music
Behavioral: Binaural beats — Binaural beats are defined as the sound that is born when two sounds of constant intensity but different frequencies are presented to both ears separately. The resultant sound perceived in the brain has a single tone and a frequency equivalent to the difference between the frequencies of the carrier sounds
  Other Names: Binaural tones
  Arms: Binaural Beats
Behavioral: White noise — White noise is a type of random sound characterized by equal intensity across all frequencies within the audible range, resulting in a steady, uniform sound similar to the static from a television or radio tuned to an unused frequency.
  Other Names: White static
  Arms: Control

SUMMARY:
Many patients suffer from dental anxiety and don't go to dentists for regular checkups. This can lead to the initiation and progression of dental caries, which, if not controlled at the right time, can lead to the loss of the tooth itself. Many forms of distraction have been used to overcome this; music is also one of them. The main objective of this study is to compare the effectiveness of binaural beats and 432 Hz music in reducing preoperative dental unease and anxiety among adult patients undergoing root canal treatment in a dental teaching hospital. The null hypothesis is that both binaural beats and 432 Hz-frequency music are not effective in reducing preoperative dental anxiety among patients undergoing routine endodontic therapy in a dental teaching hospital. A total of three groups will be a part of this study, with a total sample size of 99 participants (33 participants in each group). Group A will listen to 432 Hz music for 10 minutes before the procedure, Group B will listen to binaural beats for 10 minutes before the procedure; and Group C (active control group) will listen to white noise for 10 minutes before the procedure. The Visual Analog Scale for Anxiety will be used to assess the anxiety levels before local anesthesia administration, after local anesthesia administration, and 10 minutes after listening to sounds. Then root canal treatment will be completed as a routine procedure.

DETAILED DESCRIPTION:
i. Background Patients undergoing routine endodontic treatment often encounter severe preoperative and intraoperative anxiety that can increase the perception of pain intensity and decrease patient's cooperation with the dentist. Many audio distraction techniques have been used as a non-pharmacological means of anxiety reduction in dentistry for the past few years, and they have shown great results.

ii. Objective The main objective of this study is to compare the effectiveness of binaural beats and 432 Hz music in reducing preoperative dental unease and anxiety among adult patients undergoing routine, nonsurgical endodontic treatment in dental teaching hospital.

iii. Methodology In this randomized controlled clinical trial, a total of 99 adult patients will be recruited and will be randomly divided into three groups based on the anxiety reduction method. The first group (n = 33) will listen to music tuned to 432 Hz using wireless headphones. The second group (n = 33) will listen to binaural beats using wireless headphones, and the third group (n = 33), the control group, will listen to white noise using wireless headphones. All the patients will be informed about the procedure, and anxiety will be measured using the Visual Analogue Scale before the administration of local anesthesia. After the administration of local anesthesia, a second measurement of anxiety level will be recorded. After that, the group A will be asked to listen to 432 Hz audios using wireless headphones, group B will be requested to listen to binaural sounds using wireless headphones, and the group C (active control group) will listen to white noise using wireless headphones. After 10 minutes, anxiety will be measured again using the Visual Analog Scale. The root canal treatment will be completed in the usual way.

vi: Sequence Generation: Participants will be randomized using a lottery method to either one of the interventional groups or the control group. This method will ensure that each participant has an equal chance of being assigned to either group. 99 small pieces of paper will be made; 33 of them will have the letter 'A' written on them, 33 of them will have the letter 'B' written on them, and the remaining 33 will have the letter 'C' written on them, denoting their respective groups. All of these chits will be folded four times and placed in a hat. The participants will be asked to draw one piece of paper from the hat to be assigned to one group.

vii: Blinding: The participants and outcome assessors will be blinded in this research (double blinded). The participants will not know about their group assignment or the intervention they will receive and the outcome assessors will not know about what intervention has been given to the patients.

viii: Allocation Concealment: The lottery draw will be conducted by an independent person not involved in the study to ensure allocation concealment.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients.
* Patients between the age group of 18-45 years.
* Patients who are appointed for endodontic treatment.
* Maxillary or mandibular teeth with a history of pulp necrosis or no history of preoperative pain.

Exclusion Criteria:

* Patients who will require emergency dental treatment.
* Patients who will be taking antidepressants or medications for any kind of disease.
* Patients who will have any kind of hearing impairment.
* Patients who will be suffering from any kind of chronic, systemic, endocrine, or mental disease.
* Pregnant or lactating women and pediatric patients.
* Smokers.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Change in Pre-operative Dental Anxiety score using Visual Analog Scale for Anxiety | 10 minutes after the sound intervention
  The visual analog scale for anxiety is a 100-mm horizontal line portrayed on paper, with the left side of the line depicting "no anxiety" and the right side of the line depicting "worst anxiety imaginable," with written instructions of marking a point on the line matching the anxiety level of the patients. The closer the mark will be from the left point of no pain, the more successful the intervention will be.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Hafsa Zaki, Principal Investigator — DUHS
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
There is some information that can be sensitive to some patients. Sharing this data can compromise their confidentiality and cause a breach of their privacy. Anonymous data can be shared upon request.

REFERENCES:
- [Background] Karapicak E, Dulger K, Sahin E, Alver A. Investigation of the effect of music listened to by patients with moderate dental anxiety during restoration of posterior occlusal dental caries. Clin Oral Investig. 2023 Jul;27(7):3521-3530. doi: 10.1007/s00784-023-04966-8. Epub 2023 Mar 24. PMID 36959385
- [Background] Menziletoglu D, Guler AY, Cayir T, Isik BK. Binaural beats or 432 Hz music? which method is more effective for reducing preoperative dental anxiety? Med Oral Patol Oral Cir Bucal. 2021 Jan 1;26(1):e97-e101. doi: 10.4317/medoral.24051. PMID 33247575
- [Background] Dabiri R, Monazzam Esmaielpour MR, Salmani Nodoushan M, Khaneshenas F, Zakerian SA. The effect of auditory stimulation using delta binaural beat for a better sleep and post-sleep mood: A pilot study. Digit Health. 2022 May 20;8:20552076221102243. doi: 10.1177/20552076221102243. eCollection 2022 Jan-Dec. PMID 35615269
- [Background] Di Nasso L, Nizzardo A, Pace R, Pierleoni F, Pagavino G, Giuliani V. Influences of 432 Hz Music on the Perception of Anxiety during Endodontic Treatment: A Randomized Controlled Clinical Trial. J Endod. 2016 Sep;42(9):1338-43. doi: 10.1016/j.joen.2016.05.015. Epub 2016 Jul 16. PMID 27430941
- [Background] Calamassi D, Li Vigni ML, Fumagalli C, Gheri F, Pomponi GP, Bambi S. The Listening to music tuned to 440 Hz versus 432 Hz to reduce anxiety and stress in emergency nurses during the COVID-19 pandemic: a double-blind, randomized controlled pilot study. Acta Biomed. 2022 May 12;93(S2):e2022149. doi: 10.23750/abm.v93iS2.12915. PMID 35545982
- [Background] Aravena PC, Almonacid C, Mancilla MI. Effect of music at 432 Hz and 440 Hz on dental anxiety and salivary cortisol levels in patients undergoing tooth extraction: a randomized clinical trial. J Appl Oral Sci. 2020;28:e20190601. doi: 10.1590/1678-7757-2019-0601. Epub 2020 May 11. PMID 32401941
- [Background] Isik BK, Esen A, Buyukerkmen B, Kilinc A, Menziletoglu D. Effectiveness of binaural beats in reducing preoperative dental anxiety. Br J Oral Maxillofac Surg. 2017 Jul;55(6):571-574. doi: 10.1016/j.bjoms.2017.02.014. Epub 2017 Mar 18. PMID 28325532
- [Derived] Zaki H, Ahmed S, Rehman Qazi FU, Fatima N, Ali YS. Comparing binaural beats and 432 Hz music for reduction of preoperative anxiety in root canal patients: a randomized controlled trial. J Pak Med Assoc. 2025 Apr;75(4):540-544. doi: 10.47391/JPMA.21023. PMID 40269359